CLINICAL TRIAL: NCT02520765
Title: Obesity Index That Better Predict Ovarian Response: Body Mass Index, Waist Circumference, Waist Hip Ratio, or Waist Height Ratio in Women Undergoing ICSI
Brief Title: Obesity Index That Better Predict Ovarian Response
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed El Kotb Abdel Fattah, Doctor, Ain Shams University
Other Study IDs: obesity index in ICSI
Record Dates: First submitted 2015-08-02; First posted 2015-08-13 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Infertility
Keywords: Obesity Index, ICSI
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is designed to assess the accuracy of Body Mass Index ,Waist Circumference ,Waist Hip Ratio or Waist Height Ratio as a predictor of ovarian response in women undergoing ICSI.

DETAILED DESCRIPTION:
Obesity is an increasingly serious health concern worldwide, and its association with many diseases has been demonstrated. Obesity as it relates to infertility is also being studied All these studies used body mass index (BMI) to determine obesity. Although it is the most commonly used parameter to measure obesity, BMI does not provide an accurate measure of a person's body composition, including body fat.

Almost all studies conducted on this subject used body mass index (BMI) as the measure of obesity; however, using only BMI might be the wrong strategy. Interestingly, some studies on the cardiovascular system found protective effects of BMI and as a result a new term, 'obesity paradox,' emerged. Later studies used waist-to-hip (W/H) ratio and wrist circumference (WC) as a measure of obesity, and showed the exact effect of body fat distribution and obesity on the cardiovascular system

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for ICSI

Exclusion Criteria:

* Poor Responders.
* Poly cystic ovary syndrome.
* Previous ovarian surgeries.
* Patients with ovarian cysts
* patients with endometriosis
* women age more than 35 years

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 200 patients who are admitted to the IVF center at Ain Shmas University hospital and scheduled for ICSI
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-08 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
number of oocytes | 1 month
  number f oocytes counted at the oocyte retrieval day during ICSI

SECONDARY OUTCOMES:
clinical pregnancy rate | 7 Weeks
  detection of fetal cardiac activity by transvaginal ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed dr kotb, MD, Principal Investigator — Ain Shams University
Locations (1):
- Faculty of Medicine, Ain Shams University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No